CLINICAL TRIAL: NCT06944730
Title: Trunk and Lower Limb Movement Quality and Stability Improvement in People With Chronic Low Back Pain Following Different Types of Isometric Trunk Muscle Training
Brief Title: Movement Quality and Balance Improvement in People With Chronic Low Back Pain Following Trunk Muscle Training
Acronym: CLBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, SUTANTO Dhananjaya, Post-Doctorate Fellow, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HongKongPU RS; 2022.176 (Other: CUHK-NTEC CREC)
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: movement quality; balance; trunk muscle training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Structural Exercise (Experimental): Single armed dumbbell row, push up and single legged deadlift exercises, done three times per week for eight weeks
  Interventions: Behavioral: Structural Exercise
- Isolated Trunk Exercise (Experimental): Plank, side bridge, and bird dog isometric holds, done three times per week over eight weeks training
  Interventions: Behavioral: Isolated Trunk Exercise
- Control (Sham Comparator): Back school education where participants are taught about healthy seating position, how to carry loads, and maintaining an active daily lifestyle.
  Interventions: Behavioral: Back school

INTERVENTIONS:
Behavioral: Structural Exercise — Multi-joint limb movement with force vector through the spine. The spine is held at neutral position
  Arms: Structural Exercise
Behavioral: Isolated Trunk Exercise — Holding the spine in neutral position with no limb movement, with static loading through the spine
  Arms: Isolated Trunk Exercise
Behavioral: Back school — Patient education that has been proven to not be effective and has been used as control in past low back pain intervention studies
  Arms: Control

SUMMARY:
The goal of this project is to assess if Chronic Low Back Pain (CLBP) participant's movement quality and balance variables can change after training that decreases their pain and disability. It will also compare the difference between structural exercise (SE) and isolated trunk exercise (ITE). The main questions it aims to answer are:

1. What are the effect of the training on the participant's movement quality and balance.
2. What are the difference between different types of trunk muscle training on people with CLBP.

Researchers will compare SE, ITE and control. Control group will receive back school education that was shown not to be effective in reducing pain and disability.

Participants will:

1. Do home and in-lab based SE or ITE training, or maintain active daily living over 2 months.
2. Complete the pain and disability questionnaire and do several physical functioning tests while having their trunk and lower limb movement and muscle activation measured.

DETAILED DESCRIPTION:
Both ITE and SE training are equalized in terms of training intensity based on rate of perceived exertion, training duration per session, training frequency, and intervention period. Training intensity measurement does not use other methods of quantification as ITE training does not increase heart rate or blood lactate significantly regardless of the intensity.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) 18-25 kg/m2
* experiencing intermittent pain lasting at least 3 months
* had Oswestry Disability Index (ODI) score ranging between 17% and 45%.

Exclusion Criteria:

* exercise contraindication based on physical activity readiness questionnaire
* indication or diagnosis of other chronic diseases (such as cancer, cardiovascular disease, diabetes, bone fracture, or infection)
* artificial lower limb joints, history of spinal surgery, walking aid use
* personal mobility restrictions (due to connective tissue diseases, rheumatoid arthritis, or central nervous system disorders)
* pregnancy or within 1 year post partum

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Lower lumbar active range of motion | Same day as first day of intervention and within one week after intervention
  active range of motion of the lower lumbar area during five-repetitions sit-to-stand test.
Segmental movement coordination | Same day as first day of intervention and within one week after intervention
  Lumbar-to-pelvis and pelvis-to-femur movement coordination as quantified by mean absolute relative phase angle during five-repetitions sit-to-stand. Smaller number indicates greater coordination between the two segments.
Segmental movement stability | Same day as first day of intervention and within one week after intervention
  lumbar-to-pelvis and pelvis-to-femur movement stability as quantified by deviation phase during five-repetitions sit-to-stand. Greater number indicates lesser segmental movement stability.
Postural stability | Same day as first day of intervention and within one week after intervention
  Center-of-pressure normalized mean velocity during Y-balance test. Smaller number indicate greater stability
Postural Control | Same day as first day of intervention and within one week after intervention
  normalized leg reach during y-balance test, with larger number indicating greater postural control.
Perceived pain | Same day as first day of intervention and within one week after intervention
  score from numerical pain rating scale from zero (0) to ten (10), with 0 indicating no pain.
Perceived disability | Same day as first day of intervention and within one week after intervention
  Score based on oswestry disability index scoring from zero (0) to one hundred (100) percent, with zero indicating no disability.
5RSTS time | Same day as first day of intervention and within one week after intervention
  Time required to complete five-repetitions sit-to-stand with smaller time indicating better performance.

SECONDARY OUTCOMES:
LAP performance | Same day as first day of intervention and within one week after intervention
  time required to complete the lift and place test with lesser time indicating greater performance
Muscle synergy | Same day as first day of intervention and within one week after intervention
  Muscle synergy as measured by the surface electromyography (SEMG) output of the latissimus dorsi, longissimus pars thoracis, longissimus pars lumborum, external oblique, rectus abdominis, gluteus maximus and biceps femoris muscle both on left and right side during all functional tests. SEMG signals would then be processed using non-negative matrix factorization to find the underlying muscle synergies

CONTACTS AND LOCATIONS:
Overall Officials: Billy CL So, Prof., Study Director — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant pre and post outcome measures along with anonymized individual participant demographic data
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: a proposal that describes planned analyses must be submitted to primary investigator, and once agreed, data sharing agreement would then signed prior to data sharing.
URL: https://libguides.lb.polyu.edu.hk/prdr/restrictedaccess

REFERENCES:
- [Background] Sutanto D, Ho CY, Wong SHS, Pranata A, Yang Y. Difference in movement coordination and variability during Five-Repetition Sit-to-Stand between people with and without Chronic Low back pain. J Biomech. 2025 Mar;181:112531. doi: 10.1016/j.jbiomech.2025.112531. Epub 2025 Jan 19. PMID 39855104
- [Background] Sutanto D, Yang YJ, Wong SH. A novel physical functioning test to complement subjective questionnaires in chronic low back pain assessments. Spine J. 2023 Apr;23(4):558-570. doi: 10.1016/j.spinee.2022.12.008. Epub 2022 Dec 17. PMID 36535534
- [Background] Panjabi MM. The stabilizing system of the spine. Part I. Function, dysfunction, adaptation, and enhancement. J Spinal Disord. 1992 Dec;5(4):383-9; discussion 397. doi: 10.1097/00002517-199212000-00001. PMID 1490034
- [Background] Sutanto D, Ho RST, Poon ETC, Yang Y, Wong SHS. Effects of Different Trunk Training Methods for Chronic Low Back Pain: A Meta-Analysis. Int J Environ Res Public Health. 2022 Mar 1;19(5):2863. doi: 10.3390/ijerph19052863. PMID 35270557
- [Background] Chiarotto A, Boers M, Deyo RA, Buchbinder R, Corbin TP, Costa LOP, Foster NE, Grotle M, Koes BW, Kovacs FM, Lin CC, Maher CG, Pearson AM, Peul WC, Schoene ML, Turk DC, van Tulder MW, Terwee CB, Ostelo RW. Core outcome measurement instruments for clinical trials in nonspecific low back pain. Pain. 2018 Mar;159(3):481-495. doi: 10.1097/j.pain.0000000000001117. PMID 29194127